CLINICAL TRIAL: NCT06028087
Title: Real-World Mapping Antithrombotic Regimens in Multiple Myeloma Patients on Treatment (The MAMMOTH Study of the GIMEMA Working Party on Hemostasis and Thrombosis)
Brief Title: Real-World Mapping Antithrombotic Regimens in MM Patients on Treatment
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ET0123
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma; Diagnosis
MeSH Terms: conditions — Multiple Myeloma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about antithrombotic regimens in Multiple myeloma patients. The main question it aims to answer is the efficacy of different types of thromboprophylaxis (antiplatelet agents, heparins, oral anticoagulants) in preventing venous thromboembolism (VTE).

DETAILED DESCRIPTION:
This is an observational prospective cohort study aimed at assessing the efficacy of different types of thromboprophylaxis in MM patients; the setting is the GIMEMA network of the Italian haematological Centers.

The observation time for each patient will be of 3 years from the start of the active treatment for MM. Patients will remain in the study regardless of the stage of disease, type of treatment (induction, transplantation, maintenance), type of antithrombotic prophylaxis, occurrence of thrombosis.

Four cohorts will be identified: cohort 1 will include patients without thromboprophylaxis, cohort 2 will include patients receiving antiplatelet agents, cohort 3 will include patients receiving heparins, and cohort 4 will include patients receiving oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years of age.
2. New diagnosis of symptomatic MM according to the CRAB or the SLIM criteria of the International Myeloma Working Group
3. First active treatment for MM started after recruitment in the study
4. Signed informed consent

Exclusion Criteria:

1. Patients having had thrombosis within 6 months before diagnosis of MM
2. Patients with need of combined antithrombotic regimens (i.e. VKA or DOAC or LMWK and one or two antiplatelet drugs)
3. Ongoing first active treatment for MM initiated before the starting of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a newly diagnosis of symptomatic Multiple myeloma treated at the Italian haematological Centers of the GIMEMA network. Patients will be enrolled prior to any treatment for MM.
Sampling Method: Non-Probability Sample
Enrollment: 736 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Rate of venous thromboembolism according to different thromboprophylaxis strategies | 3 years
  Efficacy of different thromboprophylaxis strategies vs no thromboprophylaxis in terms of rate of VTE in patients newly diagnosed:
  1. Comparison of VTE rate in patients treated with antiplatelet agents vs no thromboprophylaxis
  2. Comparison of VTE rate in patients treated with heparins vs no thromboprophylaxis
  3. Comparison of VTE rate in patients treated with oral anticoagulants vs no thromboprophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Valerio De Stefano, Principal Investigator — Università Cattolica, Fondazione Policlinico A. Gemelli IRCCS, Roma
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS UOC Servizio e DH di Ematologia, Roma, Italy

IPD SHARING:
Plan to Share IPD: No